CLINICAL TRIAL: NCT06444477
Title: Molecular Analysis of Thrombocytopenia and Cancer (MATAC): Investigating Antigenic Mimicry Between Platelets and Tumor Cells in Patients With Immune Thrombocytopenia (ITP) Associated With Cancer
Acronym: MATAC
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2024/16
Record Dates: First submitted 2024-05-14; First posted 2024-06-05 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Immune Thrombocytopenia; Immune Thrombocytopenic Purpura; Neoplasms; Cancer
Keywords: Proteomics; Mortality; Side Effects; Multicenter; Retrospective
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Neoplasms | interventions — Inosine Triphosphate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a definite diagnosis of both ITP and cancer
  Interventions: Other: ITP and cancer

INTERVENTIONS:
Other: ITP and cancer — ITP and cancer

SUMMARY:
The association between hematologic malignancies and ITP is well described, but this link is much less clear with solid cancers. In cases of ITP associated with cancers, specific cancer treatment can lead to remission or even cure of ITP. Thus, our hypothesis was that chronic expression of GPIIB by tumor cells could have initiated an autoimmune loop against GPIIB, leading to the onset and perpetuation of ITP.

DETAILED DESCRIPTION:
Autoimmune thrombocytopenia, also known as immune thrombocytopenic purpura (ITP), is a rare autoimmune disease characterized by platelet destruction and impaired production, posing a life-threatening risk due to bleeding complications. The pathophysiology of ITP involves complex mechanisms, including both defective platelet production and auto-reactivity of B and T lymphocytes leading to the production of autoantibodies against platelets, found in 35 to 55% of cases. Additionally, in the context of neoplasia, some patients may develop varying degrees of thrombocytopenia, exacerbating morbidity and mortality. A multicenter, retrospective study will collect data from routine care, including birth date, gender, biological parameters related to ITP, dates of treatment initiation and diagnosis of ITP and cancer, types of treatments, and outcomes such as survival or death, without additional medical interventions or appointments.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a definite diagnosis of both ITP and cancer;
* Synchronous diagnosis of ITP and cancer;
* Onset of ITP occurring 6 months before or after the diagnosis of cancer.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a definite diagnosis of both ITP and cancer
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Remission rate of ITP at 6 months after specific cancer treatment | At baseline (Day 0)

SECONDARY OUTCOMES:
All-cause mortality | At baseline (Day 0)
Side effects related to ITP and its treatment | At baseline (Day 0)
Side effects related to its treatment | At baseline (Day 0)
Clinical description of the characteristics of ITP associated with a diagnosis of solid cancer | At baseline (Day 0)
Biological description of the characteristics of ITP associated with a diagnosis of solid cancer | At baseline (Day 0)
Demographic description of the characteristics of ITP associated with a diagnosis of solid cance | At baseline (Day 0)
Therapeutic description of the characteristics of ITP associated with a diagnosis of solid cance | At baseline (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Etienne RIVIERE, MD, Principal Investigator — University Hospital, Bordeaux
Locations (20):
- France (20):
  - AP-HP Hôpital Jean Verdier service de médecine interne, Bondy
  - CHU de Clermont-Ferrand - service de médecine interne, Clermont-Ferrand
  - AP-HP Hôpital Mondor service de médecine interne, Créteil
  - AP-HP Hôpital Bicêtre service de médecine interne, Le Kremlin-Bicêtre
  - CHU de Lille - service d'Hématologie, Lille
  - HCL - service d'Hématologie, Lyon
  - AP-HM Hôpital la Timone - service de médecine interne, Marseille
  - CHU de Montpellier - service d'Hématologie, Montpellier
  - CHRU de Nancy - service de Médecine Interne et Immunologie Clinique, Nancy
  - CHU de Nantes - service de médecine interne, Nantes
  - CHRU d'Orléans - service de Médecine interne, Orléans
  - CHRU d'Orléans - service de réanimation, Orléans
  - AP-HP Hôpital Bichat service de médecine interne, Paris
  - AP-HP Hôpital Saint-Antoine service de médecine interne, Paris
  - AP-HP Hôpital Saint-Louis service immuno-hématologie, Paris
  - CHU de Bordeaux Service de Médecine Interne et Maladies Infectieuses, Pessac
  - CHU de Poitiers - service de médecine interne, Poitiers
  - CHRU de Strasbourg - service de médecine interne, Strasbourg
  - CHU de Toulouse - service de médecine interne, Toulouse
  - CHU de Tours - service de médecine interne, Tours